CLINICAL TRIAL: NCT03729817
Title: VERiTAS-2 REFRESH ICAS (REstoring Flow by REvascularization With Submaximal Angioplasty in Hemodynamic IntraCranial Atherosclerotic Stenosis)
Brief Title: REstoring Flow by REvascularization With Submaximal Angioplasty in Hemodynamic IntraCranial Atherosclerotic Stenosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Sepideh Amin-Hanjani, Professor, Vice-Chair Department of Neurosurgery, Case Western Reserve University, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023
Record Dates: First submitted 2018-10-16; First posted 2018-11-05 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Intracranial Atherosclerotic Disease; Stroke; Angioplasty, Balloon; Hemodynamics; Device Safety
Keywords: Intracranial atherosclerotic disease; Stroke; Angioplasty, Balloon; Hemodynamics; Device Safety
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Subjects will be recruited into a prospective single-arm multi-center pilot study to assess the safety of submaximal balloon angioplasty in conjunction with intensive medical therapy in patients with hemodynamically-compromised symptomatic 70-99% atherosclerotic intracranial stenosis (ICAS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Submaximal balloon angioplasty plus intensive medical therapy (Experimental): Endovascular intervention with submaximal balloon angioplasty
  Interventions: Device: Submaximal balloon angioplasty

INTERVENTIONS:
Device: Submaximal balloon angioplasty — An endovascular procedure involving inflation of a balloon catheter undersized to 50-75% of normal vessel diameter to perform angioplasty of a stenotic blood vessel segment, with the goal of increasing blood flow.

SUMMARY:
By assessing the safety and durability of an endovascular intervention, this study will justify and inform the design of a subsequent seamless feasibility/pivotal trial aimed at the treatment of intracranial atherosclerotic stenosis (ICAS), an entity which carries a high risk of stroke despite existing medical therapies, and has no other treatment options. Given the global burden of ICAS as a leading cause of stroke, there is a high potential for public health impact not just in the U.S., but world-wide.

DETAILED DESCRIPTION:
VERiTAS II REFRESH ICAS is a prospective single-arm multi-center pilot study to assess the safety of submaximal balloon angioplasty in conjunction with intensive medical therapy in patients with hemodynamically-compromised symptomatic 70-99% atherosclerotic intracranial stenosis (ICAS). This study builds on lines of evidence from prior prospective studies that established the markedly elevated risk of subsequent stroke in ICAS patients with hemodynamic compromise, and preliminary data from small case series that support submaximal angioplasty as a potentially safe option for revascularization. The primary objective of the current study is to determine the safety of submaximal balloon angioplasty for treatment of hemodynamically-compromised symptomatic ICAS. The secondary objectives are to obtain preliminary estimates for the risk of subsequent in-territory stroke at one year, to evaluate the hemodynamic effect of submaximal balloon angioplasty on distal blood flow, and to examine the hemodynamic durability of submaximal balloon angioplasty over follow-up.

A total of 159 patients will be enrolled in this open-label study to receive the submaximal angioplasty intervention in conjunction with intensive medical therapy. Patients with stroke attributable to ICAS serve as the source population for the study, and will be identified as inpatients or outpatients at participating centers or their referring sites. Patients with recently (within 30 days prior to enrollment) symptomatic 70-99% ICAS of the intracranial internal carotid (ICA), middle cerebral (MCA), vertebral (VA) or basilar (BA) artery will first be identified by a standard of care screening imaging modality (e.g. CTA, MRA, TCD). If the patient is eligible based on available inclusion/exclusion criteria, informed consent will be obtained and MRI/ quantitative magnetic resonance angiography (QMRA) will be performed (if not already as standard care); patients demonstrating evidence of hemodynamic compromise based on borderzone infarct pattern for the anterior circulation (ICA and MCA) and by low flow state on QMRA for the posterior circulation (VA and BA) will be considered eligible. QMRA will be used for determination of eligibility in posterior circulation ICAS patients, but will be performed in both anterior and posterior circulation patients as a baseline for hemodynamic comparison post-procedure. The patient will then undergo CTA (if not performed already as standard care) to confirm eligible intracranial ICAS.

The participant will undergo angiography, and upon final angiographic confirmation of eligibility will undergo submaximal angioplasty in accordance with the study protocol, followed by SAMMPRIS regimen intensive medical therapy, including initial dual antiplatelet therapy (aspirin and clopidogrel for 3 months followed by aspirin monotherapy), and targeting primary and secondary stroke risk factors. Assistance in achieving the risk factor goals will be provided by an INTERVENT lifestyle coach, who will call the participant by phone at 1, 3, 5, 7, 9, 11 weeks, and then every 4 weeks throughout follow-up. On a scheduled basis, INTERVENT will send a report of the participant's progress and goals for risk factor modification to the participant and study coordinator/ study neurologist. Participants will have follow-up for a total of one year. All participants will have clinical visits at 1, 4, 8, and 12 months, performed by local study personnel not directly involved with the angioplasty procedure. The study visits will include assessment of neurological, functional and cognitive status, as well as status of primary and secondary stroke risk factor control. QMRA will be performed post procedure and at 12 months; the follow-up QMRA results will be blinded to the local study personnel and patients. The main outcomes of interest are: (1) any periprocedural (within 30 day) stroke or death; (2) stroke in the symptomatic vessel territory; and (3) distal flow status post procedure and at follow-up (using QMRA). Additional measured endpoints will include cerebral infarct on imaging associated with temporary signs, restenosis and functional and cognitive outcomes at follow-up.

The sample size calculations have been based on a confidence interval (CI) approach aimed at determining if the intervention can be performed with a clinically specified periprocedural event rate of 5% (90% CI 2%,9%), in order to establish sufficient periprocedural safety of submaximal angioplasty to warrant further investigation in a future phase 2/3 randomized trial. The sample size calculation assumes a CI approach around the stroke/death event rate at 30 days; for the presumed event rate of 5%, a sample size of N=148 would yield a 90% CI of (2%,9%). Adjusting for the inflation factor 1.02 due to a planned interim analysis and a 5% attrition rate for the 30-day follow-up, 159 patients are required to undergo submaximal angioplasty for analysis of the primary safety endpoint. An interim analysis of safety is planned with a stopping rule if 30-day periprocedural risk exceeds 5% (i.e. lower bound of CI of observed estimate exceeds the threshold). To ensure that the intervention is stopped early if it is harmful, the timing of the interim analysis will be flexible, to occur once 30 day follow-up has been completed on one third of submaximal angioplasty patients (50 patients, accounting for attrition) or alternatively, when 13 events are observed, whichever comes first; the number of events, 13, has been specified as the minimal event number which would result in the lower bound of the 90% CI exceeding 5% and thus claim a >5% event rate. As related to the study's go/no go criteria for a future trial, our definitive no go parameter is proposed as the lower bound of the observed pre-specified CI exceeding the safety (30-day periprocedural risk) threshold of 5%. Other outcomes from the study (i.e. the secondary clinical and hemodynamic endpoints at 12 months) would also be taken into account in determining whether the procedure warrants additional study in a future seamless phase 2/3 trial.

ELIGIBILITY:
Inclusion:

* Non-severe recent stroke (within 30 days) attributed to 70-99% stenosis of intracranial artery (internal carotid, middle cerebral, vertebral, basilar); must be confirmed by CTA (or DSA if already available) for enrollment into the trial.
* Hemodynamic compromise based on borderzone infarct pattern* for the anterior circulation (internal carotid and middle cerebral artery stenosis) and by low flow state on QMRA** for the posterior circulation (vertebral and basilar artery stenosis).
* Target vessel with minimal nominal diameter of 2mm
* Target length of stenosis <18mm
* Symptoms within 30 days of enrollment
* Age ≥30 and ≤90 years old#
* Able to provide informed consent

  * *Sole or predominant borderzone infarct pattern of qualifying event, as defined by SAMMPRIS cohort analysis **Low flow state as determined by optimized flow algorithm as defined by the VERiTAS Study
  * #Those 30-49 years of age must also have the presence of established atherosclerotic disease in another vascular bed (coronary, extracranial carotid, peripheral) or the presence of 2 or more risk factors (hypertension, diabetes mellitus, hyperlipidemia, tobacco abuse within the last 2 years).

Exclusion:

* Major disabling stroke mRS >3; progressive or fluctuating deficit within 24 hours
* Hemorrhagic infarction (based on CT) within 14 days of enrollment
* Any large stroke (>5cm) to be at risk for hemorrhagic conversion
* Any neurological disease which would confound follow-up assessment
* Any co-morbid disease condition with <12 month life expectancy
* Known cardiac disease associated with elevated cardioembolic risk, specifically, atrial fibrillation, prosthetic valve, endocarditis, left atrial/ventricular thrombus, cardiomyopathy with EF<25%, cardiac myxoma
* Blood dyscrasias, specifically polycythemia vera, essential thrombocytosis, sickle cell disease
* Active bleeding diathesis, h/o major systemic hemorrhage within 30 days, active PUD, platelets<100K (severe liver impairment (AST or ALT>3 x normal, cirrhosis)
* Non-atherosclerotic stenosis including dissection, fibromuscular dysplasia, vasculitis, radiation induced vasculopathy, suspected recanalized embolus, suspected vasospastic process
* Mori C classification of stenosis (i.e. diffuse lesion, extremely angulated >90⁰, excessive proximal tortuosity) Previous treatment of target lesion with stent, angioplasty or other mechanical device
* Extracranial vertebral artery or carotid artery tortuosity, stenosis or occlusion prohibiting access to the target lesion (not exclusionary if does not prohibit access to target lesion)
* Unable or unwilling to undergo MRI
* Unable to undergo cerebral angiography
* Pregnancy
* Concurrent participation in another study which would conflict with the current study
* Allergy or contraindication to aspirin or Plavix
* Indication for warfarin or NOAC beyond enrollment (e.g. venous thrombo-embolism, atrial fibrillation)
* Thrombolytic therapy within 24 hours

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2027-10 (Estimated); Primary Completion 2031-10-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Procedural Safety | 30 days
  Any stroke (ischemic or hemorrhagic), or death, within 30 days following submaximal angioplasty

SECONDARY OUTCOMES:
Clinical Efficacy | 1 year
  Any stroke/death within 30 days or ischemic stroke in the symptomatic vessel territory at one year
Hemodynamic Success | post procedure (within 7 days)
  Initial hemodynamic effect of submaximal balloon angioplasty on treated vessel flow
Hemodynamic Durability | 1 year
  Hemodynamic durability of submaximal balloon angioplasty at follow-up in the treated vessel at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sepideh Amin-Hanjani, MD, Principal Investigator — Case Western Reserve University; Adnan Siddiqui, MD, Principal Investigator — University at Buffalo; Tanya Turan, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No